CLINICAL TRIAL: NCT01557010
Title: The Clinical Trial for Evaluation of Efficacy and Safety of DWP05195 in Postherpetic Neuralgia: Double-blind, Placebo-controlled, Randomized, Multi-center, Exploratory Clinical Trial
Brief Title: Evaluate the Efficacy and Safety of DWP05195 in Subjects With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWP05195-P003
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: DWP05195
- Treatment B (Experimental)
  Interventions: Drug: DWP05195
- Treatment C (Experimental)
  Interventions: Drug: DWP05195
- Treatment D (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: DWP05195 — Tablets, oral administration, 100mg
  Arms: Treatment A
Drug: DWP05195 — Tablets, oral administration, 200mg
  Arms: Treatment B
Drug: DWP05195 — Tablets, oral administration, 300mg
  Arms: Treatment C
Drug: Control — Tablets, oral administration, Placebo
  Arms: Treatment D

SUMMARY:
The purpose of this study is to evaluate efficacy, safety of administered DWP05195 in Postherpetic Neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects aged 20 to 80 years
* Subjects with symptoms of neuropathic pain associated with postherpetic neuralgia(PHN).
* Subjects must have pain present for > 3 months after healing of the acute herpes zoster skin rash.

Exclusion Criteria:

* Other severe pain that may potentially confound pain assessment.
* Subjects with symptoms of neuropathic pain applied Medical Equipment
* Within 2 years: Subjects were diagnosed with cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Endpoint change from the baseline after administered 8 weeks mean pain score based on the Numerical pain Rating Scale(NPRS) from the subject's daily pain diary | 8 weeks

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473